CLINICAL TRIAL: NCT04060251
Title: Is There an Alternative to Immediate Home Physical Therapy Following Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to limitations caused by COVID, enrollment targets could not be met.
Sponsor: Wolfgang Fitz, M.D. (Other)
Collaborators: CyMedica Orthopedics, Inc (Industry)
Responsible Party: Sponsor-Investigator, Wolfgang Fitz, M.D., Assistant Professor of Orthopedic Surgery, Harvard Medical School, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018P000932
Record Dates: First submitted 2019-04-03; First posted 2019-08-19 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Total Knee Arthroplasty
Keywords: Total knee arthroplasty; Physical therapy; Neuromuscular electrical stimulation; Telemedicine
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants assigned to one of three groups, there is no crossover. Participants remain in their assigned group until completion of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group 1, iGetBetter Group (Experimental): Use only iGetBetter for the 3 months preceding surgery. After surgery, you will be given a new, Post-Op program to use for 2-3 months. For the first 3 weeks, you will only use iGetBetter. After those 3 weeks, you will receive outpatient physical therapy in addition to iGetBetter, approximately twice per week for the next 6-8 weeks.
  Interventions: Other: iGetBetter telemedicine physical therapy
- Group 2, E-vive Group (Experimental): You will use iGetBetter starting 3 months out from surgery. You will receive CyMedica's electrical-stimulation garment during the preoperative appointment. In addition to iGetBetter, you will wear the conductive garment two times each day for the last 3 weeks before surgery. After surgery, for the first 3 weeks you will only use the conductive garment, and will not use iGetBetter. After those 3 weeks, you will receive outpatient physical therapy in addition to wearing the brace, approximately twice per week for the next 6-8 weeks. You will not need to return the brace after this time is up, and you may keep the brace, if you so choose, at no cost.
  Interventions: Device: CyMedica e-vive™ System; CY-1000
- Group 3, Physical Therapy Group (No Intervention): You will receive only iGetBetter for the 3 months preceding surgery. After surgery, you will receive only home physical therapy, and will not use iGetBetter. After those three weeks, you will receive outpatient physical therapy approximately twice per week for the next 6-8 weeks.

INTERVENTIONS:
Device: CyMedica e-vive™ System; CY-1000 — All the patients in Group 2 will be given the CyMedica Orthopedics e-vive system 3 weeks before the surgery. The patients will begin using the unit after their first pre-intervention measurements are taken.
  Patients will be instructed to apply the e-vive NMES Strength therapy twice a day, 5 days a week. The NMES Strength program is 20 minutes in length. Treatment intensity (adjustable from 1 to 100 in NMES programs) is required to be set at the highest tolerable limit for the patients.
  Stimulation from the garment will have the following parameters: frequency of 50 Hz; pulse duration of 5 ms; time on: 12.8 seconds; and time off: 10 seconds. The total contraction time in a 20-minute treatment will be 11 minutes. The waveform will be pulsed and asymmetrical.
  Other Names: Powered Muscle Stimulator or Neuromuscular Electrical Stimulator (NMES); IPF Transcutaneous Nerve Stimulator (TENS) for pain relief; GZJ Goniometer; KQX
  Arms: Group 2, E-vive Group
Other: iGetBetter telemedicine physical therapy — Group 1 patients will only use a Post-Op program from iGetBetter for the first 3 weeks after surgery. After those 3 weeks have elapsed, Group 1 patients will receive outpatient physical therapy in addition to iGetBetter, approximately twice per week for the next 6-8 weeks as all other groups.
  Arms: Group 1, iGetBetter Group

SUMMARY:
The purpose of this study is to evaluate how different pre-operative therapeutic approaches affect quad strength and patient satisfaction after total knee replacements. There are three treatments groups: standard physical therapy protocol, the use of CyMedica NMES garments, and a telemedical home therapy program.

DETAILED DESCRIPTION:
Patients undergoing total knee replacement (TKR) at Brigham and Women's Faulkner Hospital and meet all eligibility criteria will be informed about the study and asked if they would like to participate. The research assistant (RA) will screen upcoming surgeries and call all qualifying patients to inform them of the study. Those who show interest will be offered the opportunity to discuss with both the RA and Principal Investigator (PI). Upon agreement, the patient's consent will be obtained and they will be randomly assigned to one of three treatment groups using a computer-generated randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Owns a device with internet connection
* Can download the E-vive application for the contractile garment (has sufficiently up-to-date phone or tablet, or has family member with such a device).
* Has a rudimentary understanding of Internet technology, especially e-mail
* Has a flexion of 90 o and flexion contracture of 5 o at the point of discharge
* Approved by a physical therapist to participate safely in the study at the time of discharge

Exclusion Criteria:

* Rheumatoid arthritis
* History of epilepsy
* Implanted and body-worn electronic medical device, including cardiac pacemakers, neural stimulators, insulin pumps, etc.
* Poor understanding of the use of the brace/electrical stimulation
* Lesions on the skin over the thigh
* Uncontrolled diabetes
* Uncontrolled hypertension
* Bilateral TKA or UKA planned
* If female, pregnant
* Cannot use non-operated leg postoperatively to propel active motion splint, caused by neurological or muscular diseases such as complete or incomplete paralysis or other causes of weakness with an inability to bend or extend knee
* Loss of sensation in operated or non-operated leg
* Has below- or above-knee amputations of non-operative leg
* Below- knee amputation of operated side
* Chronic pain syndrome with inability to walk
* Taking chronic narcotics and/or is taking more than 10mg codeine per day, or any Hydrocodone, or more than 200 mg of tramadol, or any other narcotics prescribed for moderate to severe pain
* Involved in pain clinics for chronic pain, or pain that is not related to the knee
* Has been diagnosed with knee disorder other than osteoarthritis, post-traumatic osteoarthritis, gout, pseudo gout, or any inability to walk due to disorders unrelated to the knee (e.g., hip disorders, spinal stenosis, paralysis, hemi-paralysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Fitz, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Faulkner Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2, E-vive Group: You will use iGetBetter starting 3 months out from surgery. You will receive CyMedica's electrical-stimulation garment during the preoperative appointment. In addition to iGetBetter, you will wear the conductive garment two times each day for the last 3 weeks before surgery. After surgery, for the first 3 weeks you will only use the conductive garment, and will not use iGetBetter. After those 3 weeks, you will receive outpatient physical therapy in addition to wearing the brace, approximately twice per week for the next 6-8 weeks. You will not need to return the brace after this time is up, and you may keep the brace, if you so choose, at no cost.
  CyMedica e-vive™ System; CY-1000: All the patients in Group 2 will be given the CyMedica Orthopedics e-vive system 3 weeks before the surgery. The patients will begin using the unit after their first pre-intervention measurements are taken.
  Patients will be instructed to apply the e-vive NMES Strength therapy twice a day, 5 days a week. The NMES Strength program is 20 minutes in length. Treatment intensity (adjustable from 1 to 100 in NMES programs) is required to be set at the highest tolerable limit for the patients.
  Stimulation from the garment will have the following parameters: frequency of 50 Hz; pulse duration of 5 ms; time on: 12.8 seconds; and time off: 10 seconds. The total contraction time in a 20-minute treatment will be 11 minutes. The waveform will be pulsed and asymmetrical.
Period: Overall Study
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Started | 8 (Due to limitations caused by COVID, enrollment targets could not be met.) | 6 (Due to limitations caused by COVID, enrollment targets could not be met.) | 7 (Due to limitations caused by COVID, enrollment targets could not be met.)
Completed | 0 (Due to limitations caused by COVID, enrollment targets could not be met.) | 0 (Due to limitations caused by COVID, enrollment targets could not be met.) | 0 (Due to limitations caused by COVID, enrollment targets could not be met.)
Not Completed | 8 | 6 | 7
Not completed — Study terminated due to low enrollment. | 7 | 5 | 7
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Due to limitations caused by COVID, enrollment targets could not be met. Data was not collected for targets that were enrolled. No analysis of population was performed because no data was collected and therefore cannot be reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Sit-to-stand Time
Description: Change in sit-to-stand capabilities
Time Frame: Preoperative (varies) and postoperative appointments (2 months after surgery)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Quadriceps Strength
Description: Change in quadriceps strength in lbs of force, as measured by PT dynamometer
Time Frame: Preoperative and postoperative appointments (2 months after surgery)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: 2 Minute Walking Time
Description: Change in distance walked in 2 minutes
Time Frame: Preoperative and postoperative appointments (2 months after surgery)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Walking Speed
Description: Change in walking speed
Time Frame: Preoperative and postoperative appointments (2 months after surgery)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: Balancing
Description: Change in proprioception (balance) as measured by 30-second single limb stance PT test
Time Frame: Preoperative and postoperative appointments (2 months after surgery)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Visual Analogue Scale (VAS) Pain
Description: Change in Visual Analog Scale for pain (1-10) 1 no pain 10 worse
Time Frame: first postoperative months (from days post-op through 2-month post-operative appointment)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Visual Analogue Scale (VAS) Nausea
Description: Change in VAS nausea (Visual Analog Scale for nausea (1-10) 1 no nausea 10 worse nausea )
Time Frame: first postoperative months (from days post-op through 2-month post-operative appointment)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Visual Analogue Scale (VAS) Satisfaction
Description: Change in VAS satisfaction (Visual Analog Scale for satisfaction (1-10) 1 not satisfied, 10 totally unsatisfied)
Time Frame: first postoperative months (from days post-op through 2-month post-operative appointment)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Readmission Rate
Description: major complication
Time Frame: Noted by PI at 2nd postoperative appointment (about 10 weeks after surgery)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Infection Rate
Description: superficial and deep infection
Time Frame: Noted by PI at 2nd postoperative appointment (about 10 weeks after surgery)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Cost Per Treatment Regimen (iGetBetter vs. CyMedica E-vive vs. Home PT)
Description: We will calculate the total cost of each treatment modality
Time Frame: Completion of study (anticipate one year from start data 4/4/2019)
Population: as for baseline characteristics
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 148 days (21.14 weeks)
Arm/Group | Group 1, iGetBetter Group | Group 2, E-vive Group | Group 3, Physical Therapy Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 1/6 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1, iGetBetter Group (N=8) | Group 2, E-vive Group (N=6) | Group 3, Physical Therapy Group (N=7)
Advanced Home PT Required (General disorders) | 1 (1) | 1 (1) | 0 (0) — Subject was determined to require more advanced home physical therapy.

LIMITATIONS AND CAVEATS:
Due to limitations caused by COVID, enrollment targets could not be met. Data was not collected for targets that were enrolled. No analysis of population was performed because no data was collected and therefore cannot be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT04060251/Prot_SAP_000.pdf